CLINICAL TRIAL: NCT04062344
Title: Acquisition of Resistant Enterobacteria During Oral Drug Challenge for Betalactams in Children
Acronym: ARET
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190252; 2019-A00755-52 (Other: IDRCB number)
Record Dates: First submitted 2019-08-19; First posted 2019-08-20 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Betalactams Hypersensitivity
Keywords: Betalactams hypersensitivity; Children; Drug provocation testing; Bacterial resistances

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Short oral drug provocation test: Minors performing a short (1-4 days) drug provocation test
  Interventions: Other: Swab
- Prolonged oral drug provocation test: Minors performing a prolonged (5-8 days)drug provocation test
  Interventions: Other: Swab

INTERVENTIONS:
Other: Swab — Rectal swab before and after the drug provocation testing
  Other Names: Rectal swab

SUMMARY:
Direct drug provocation testing, without prior skin or in vitro testing, is the reference standard for confirming the diagnosis of drug hypersensitivity reactions in children reporting mild and delayed-onset reactions. However, optimal protocol(s) have not been standardized. Although a 2-days' provocation testing protocol is effective, increasing its duration (up to 14 days) may improve its diagnosis performance without increasing the risk of severe reactions. However, a prolonged provocation testing could increase the risk of emergence of bacterial resistances in the digestive flora. Longer duration could be associated with the emergence of extended-spectrum betalactamase producing enterobacteria. However, this point has never been confirmed.

The study will include children (0-18 years); referring for histories of mild and delayed-onset reactions to betalactams. drug provocation testing will be performed with the suspected BLs in our department, as in clinical practice. Two groups of patients will be compared: a group performing short provocation testing (arbitrary defined as lasting 1 to 4 days) and a group with prolonged drug provocation testing (arbitrary defined as lasting 5-8 days). A rectal swab will be collected for each patient before the provocation testing, a second one at the end of the provocation testing. Each sample will be analyzed to detect the presence extended-spectrum betalactamase -producing enterobacteria.

DETAILED DESCRIPTION:
Drug hypersentivity in children is suspected in up to 10% of parents. However, drug hypersensitivity is rarely confirmed: its prevalence in children is estimated to be less than 0.5%. The most frequently suspected drugs are betalactams such as amoxicillin and oral cephalosporins (cefpodoxime, cefixime, cefuroxime). Most reported drug hypersensitivity reactions to betalactams in children are mild and delayed-onset, typically starting more than one hour after the first dose. These reactions often include urticaria, maculo-papular rashes, and/or edema. Amoxicillin is indicated as a first-line therapy in the majority of common infections in children. Suspicion of betalactams hypersensitivity is associated with the prescription of alternate antibiotics often less effective and that may increase the risk of bacterial resistance, morbidity and health costs. Therefore it is necessary to confirm or exclude a true betalactams hypersensitivity.

Direct drug provocation testing without prior skin or in vitro testing, is the reference standard for confirming the diagnosis of drug hypersensitivity reactions in children reporting mild and delayed-onset reactions. However, optimal protocol(s) have not been standardized. Although a 2-days' drug provocation testing protocol is effective, increasing its duration (up to 14 days) may improve its diagnosis performance without increasing the risk of severe reactions. However, a prolonged drug provocation testing could increase the risk of emergence of bacterial resistances in the digestive flora. Longer duration could be associated with the emergence of extended-spectrum betalactamase producing enterobacteria. However, this point has never been confirmed.

The aim of this study is to determine whether the risk of emergence of ESBL-producing bacteria in the digestive flora is higher in case of prolonged drug provocation testing.

Our hypothesis is that the acquisition rate of extended-spectrum betalactamase -producing enterobacteria will be higher in prolonged drug provocation testing.

As previously published, in the Pediatric Pulmonology and Allergy Department of the Necker Hospital, we perform direct drug provocation testing with the culprit drug in children with histories of mild delayed-onset reactions. Drug provocation testing is prolonged at home at normal therapeutic doses. The duration of the drug provocation testing is 1-2 days more than the chronology of the index reactions, with a maximum of eight days.

The study will include children (0-18 years), referring for histories of mild and delayed-onset reactions to betalactams. drug provocation testing will be performed with the suspected betalactam in our department, as in clinical practice. Two groups of patients will be compared: a group performing short drug provocation testing (arbitrary defined as lasting 1 to 4 days) and a group with prolonged drug provocation testing (arbitrary defined as lasting 5-8 days). A rectal swab will be collected for each patient before the drug provocation testing, a second one at the end of the drug provocation testing. Each sample will be analyzed to detect the presence extended-spectrum betalactamase -producing enterobacteria.

ELIGIBILITY:
Inclusion Criteria :

* Minors aged 0 to 18
* Consultation in Necker for an oral drug provocation test to explore mild (urticaria, edema, maculo-papulous exanthema) delayed-onset reaction (1 hour after initiation of treatment) to betalactams (amoxicillin +/-clavulanic acid, cefpodoxime, cefixime, cefuroxime)

Exclusion Criteria :

* Minors with potentially severe delayed-onset reactions (painful skin lesions, atypical target lesions, erosions of mucosa, centro facial oedema, purpuric infiltrated papules) or severe (Lyell/Stevens Johnson Syndrome, fixed drug eruption, acute generalized exanthematous pustulosis, skin rash with systemic and hypereosinophilic disorders)
* Antibiotic treatment within the past month before the drug provocation test
* Travel abroad within the past 6 months before the drug provocation test
* Cardio-respiratory failure, renal failure, hepatic impairment or any other severe chronic pathology

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minors in consultation at Necker Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-23 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Acquisition of at least one strain of extended-spectrum betalactamase-producing enterobacteria | 24 months
  Bacteriological culture with gram-negative bacteria-specific agar. Bacterial colonies will be identified by mass spectrometry (Matrix Assisted Laser Desorption Ionization technique - Time of Flight, MALDI-TOF).
  Antibiogram.

SECONDARY OUTCOMES:
Acquisition of at least one strain of third generation cephalosporin-resistant gram-negative bacteria | 24 months
  Bacteriological culture with gram-negative bacteria-specific agar supplemented with third-generation cephalosporins.
  Bacterial colonies will be identified by mass spectrometry (Matrix Assisted Laser Desorption Ionization technique - Time of Flight, MALDI-TOF).
  Antibiogram.
Metagenomic analysis of intestinal microbiota | 24 months
  Metagenomic analysis will be performed by high-throughout sequencing using next-generation high-throughout DNA sequencing technologies.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Lezmi, Doctor (PHU), Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, Paris, France